CLINICAL TRIAL: NCT05721391
Title: To Study the Impact of Frailty on Postoperative Complications in Oncosurgeries
Brief Title: Impact of Frailty on Postoperative Complications in Oncosurgery
Acronym: Frailty
Status: Completed | Type: Observational
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr Anita Kulkarni, Principal investigator, Rajiv Gandhi Cancer Institute & Research Center, India
Other Study IDs: RGCI Frailty
Record Dates: First submitted 2023-01-28; First posted 2023-02-10 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Frailty; Postoperative Complications
MeSH Terms: conditions — Frailty; Postoperative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non Frail Group: The patients in no frail group did not have any component of Frailty criteria
- Pre Frail Group: The patients in prefrail Group had 1-2 component of Frailty criteria.
- Frail Group: The patients in Frail Group had 3-5 component of Frailty criteria.

SUMMARY:
Advanced ageing is accompanied by loss of reserve in multiple organ systems leading to increased risk of complications after surgery.Frailty is a functional syndrome involving reduced physiological reserve and 25-56% of all elderly surgical patients are reported to be frail .

DETAILED DESCRIPTION:
Patients above 65 years age undergoing major Oncosurgery under general anaesthesia with or without Epidural will included , written informed consent will be obtained from all patients. Age, Heigth , Weigth , polypharmacy , smoking status , history of Diabetes ,Hypertension will be noted. Basic investigation Hb% , Serum Albumin , Serum creatinine will be done. ASA Physical status and Surgical risk will be noted .Patients will be evaluated for Frieds 5 point Frailty Assessment Scale (i) Unintended weigth loss of > 5kg in last one year.(ii) self reported exhaustion, (iii) muscle weakness (grip strength) (iv)slow walking speed,(v) Low physical activity and assigned to either No Frail Group (0 criteria) , Pre-Frail (1-2 positive criteria ), Frail (3-5 positive criteria Group).The assessment will be done in the preoperative anaesthesia clinic and include paper based questionnaire, hand dynamometer to measure muscle strength and walking test .

All patients will receive standard general anaesthesia along with Epidural for Abdomino-pelvic surgeries.Intraoperative monitoring 5 lead ECG, NIBP/IBP , SPO2, ETCO2, CVP(Optional),BIS will be done.After induction of anaesthesia Ultrasonography will be performed with curvilinear probe --- at the midpoint of femur anteriorly to measure Rectus Femoris muscle thickness of Right thigh , three consecutive readings will be measured and average of value noted for all patients.

At the end of surgery patient's neuromuscular block will be reversed and trachea extubated , if any patient requires ventilator support note will be made accordingly. Postoperative patients vitals and Input/Output charting will be done .Postoperative analgesia either epidural analgesia or intravenous opioids according to Institutional protocol will be given .Length of ICU Stay and any major cardiac , respiratory , Renal complications , re-exploration will be noted.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing major onco-surgey

Exclusion Criteria:

* Patient refusal to participate
* Age <65 years.
* Emergency surgery
* Pre-existing dementia
* Language barrier

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients 65 years old and above undergoing elective major onco- surgeries .
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
To study incidence of postoperative complications in frail patients | upto 7 days
  Postoperative major complications as myocardial infarction, Respiratory failure, cerebrovascular event, renal failure , re-exploration will be noted and statistically analysed.

SECONDARY OUTCOMES:
Length of ICU stay | upto 240 hours.
  Time from admission to the PACU to shifting to the ward will be noted in hours.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kulkarni, MD, Principal Investigator — Rajiv Gandhi Cancer Institute and Research Centre , Delhi , India
Locations (2):
- India (2):
  - Rajiv Gandhi Cancer Institute and Research Centre, New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Institute, Delhi